CLINICAL TRIAL: NCT01380067
Title: Phase 3 Study of a New Way for Laparoscopic Inguinal Hernia Repair in Pediatric
Brief Title: a New Way for Laparoscopic Inguinal Hernia Repair in Pediatric
Status: Completed | Type: Observational
Sponsor: The Second People's Hospital of GuangDong Province (Other)
Responsible Party: The Second People's Hospital of GuangDong Province, The Second People's Hospital of GuangDong Province
Other Study IDs: 8808
Record Dates: First submitted 2011-06-17; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-12

CONDITIONS: Complications of Surgical and Medical Care: General Terms
Keywords: Inguinal hernia; Lateral umbilicus ligament; Recurrence
MeSH Terms: conditions — Hernia, Inguinal; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: the patients were subjected laparoscopic purse-string knot for closing the internal hernia opening
- Group B: the lateral umbilicus ligament was used to cover the internal hernia opening after the laparoscopic purse-string knot

SUMMARY:
laparoscopic hernia sac high-ligation

* has a high recurrence rate laparoscopic hernia sac high-ligation and the lateral umbilicus ligament covering the hernia opening
* The investigators developed a method of laparoscopic hernia repair by applying a new concept in hernia repair. The hernia opening was tightened, and hernia opening region repaired with a lateral umbilicus ligament in a tension-free manner. This method combines the advantages of a secure repair achieved by the open method with the minimal invasiveness of the laparoscopic method. The investigators hypothesized that the lateral umbilicus ligament covering the internal hernia opening region after the laparoscopic purse-string knot would result in lower recurrence and the same operation relative complication.

DETAILED DESCRIPTION:
The primary outcome measure was the recurrence rate after surgery, and the secondary outcome measures included degree of postoperative pain, the amount of postoperative analgesia, procedural duration, number of days to recovery normal activity, surgical complications, cosmetic results, and patient satisfaction. The outcome was recorded at the outpatient visits 10 days, 6 months, 1 year, 3 years and 5 years after the surgery. The cosmetic result was scored (unsatisfactory = 0, satisfactory = 1, good = 2, and excellent = 3) by the patients or parents, the attending nurse, and the surgeon (maximum points = 9). The patient satisfaction was scored similarly (unsatisfactory = 0, satisfactory = 1, good = 2, and excellent = 3). The long axis of the testes was measured.

ELIGIBILITY:
Inclusion Criteria:

* unilateral inguinal hernia age between 2 and 17 years the absence of a history of abdominal or inguinal operations. Of the male patients, only those with completely descended testes were included.

Exclusion Criteria:

* the bilateral cases

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample size was calculated such that a 4% difference (α = 0.05) in recurrence rate at 5 years between the groups could be detected with a power of 0.9. This required a sample size of 510 patients. Considering an estimated drop-out rate of 10%, we aimed to enroll 600 patients.
Sampling Method: Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2000-01; Primary Completion 2005-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
recurrence rate | five years
  The outcome was recorded at the outpatient visits 10 days, 6 months, 1 year, 3 years and 5 years after the surgery.

SECONDARY OUTCOMES:
degree of postoperative pain | one year
  The outcome was recorded at the outpatient visits 10 days, 6 months, 1 year, 3 years and 5 years after the surgery.
patient satisfaction. | one year
  The patient satisfaction was scored similarly (unsatisfactory = 0, satisfactory = 1, good = 2, and excellent = 3). The long axis of the testes was measured.

CONTACTS AND LOCATIONS:
Overall Officials: kaiyun chen, MD, Study Chair — The Second People's Hospital of GuangDong Province